CLINICAL TRIAL: NCT03399656
Title: Broccoli Supplement Dose Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Qidong Liver Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB00008184
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 4 placebo tablets
  Interventions: Dietary Supplement: Placebo tablets
- Low Dose Avmacol (Active Comparator): 2 tablets Avmacol and 2 placebo tablets
  Interventions: Dietary Supplement: Avmacol tablets; Dietary Supplement: Placebo tablets
- High Dose Avmacol (Active Comparator): 4 Avmacol tablets
  Interventions: Dietary Supplement: Avmacol tablets

INTERVENTIONS:
Dietary Supplement: Avmacol tablets — The active components of Avmacol® are ground broccoli seeds that provide glucoraphanin and freeze-dried broccoli sprouts that provide a stabilized form of the enzyme myrosinase, which converts glucoraphanin to sulforaphane.
  Arms: High Dose Avmacol; Low Dose Avmacol
Dietary Supplement: Placebo tablets — MCC 90M Emcocel
  Arms: Low Dose Avmacol; Placebo

SUMMARY:
Do daily high (4 tablets) or intermediate (2 tablets) administration of the broccoli-based dietary supplement Avmacol® have improved bioavailability over a broccoli sprout beverage rich in sulforaphane and its biogenic precursor, glucoraphanin? The beverage formulation has been used successfully in the investigators' previous intervention studies in regions of China with high levels of air pollution to reduce the body burden of carcinogenic and toxic pollutants. The investigators seek to evaluate a more stable, less expensive formulation of a broccoli sprout preparation that can be used for disease prevention in future studies.

DETAILED DESCRIPTION:
The investigators will conduct a 3-armed placebo-controlled 16-day intervention with the dietary supplement Avmacol® to determine the bioavailability with repeated dosing of a simple tablet-based intervention in the study participants. As shown in Scheme 1, the 3 arms are: 1) 4 tablets of Avmacol® daily for 14 days; 2) 2 tablets of Avmacol® daily for 14 days together with 2 placebo tablets to maintain parity in consumption; and 3) 4 placebo tablets daily for 14 days. In addition, all participants will receive 4 placebo tablets for 2 consecutive run-in days prior to commencing intervention in the 3 distinct arms. Consecutive overnight (12-hour) urine samples will be collected during the 2-day run-in, the 14-day intervention and during a 5-day run-out period (total = 21 days). Additional day-time urine collections will be made at 2 timepoints: the day after administration of Avmacol® tablets begins and the day after the last administration of Avmacol® tablets. A blood sample will be collected at the beginning of the run-in and after the last Avmacol® dose (Day 17 for intervention groups, and for the placebo group) from each participant. The tablets will be taken before dinner each day.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 and ≤ 70 years who are residents of Qidong, China.
2. Able to provide written, informed consent.
3. Normal physical examination and medical history indicative of good general health with no history of chronic illness.
4. No hepatomegaly by clinical exam;
5. Normal liver function tests (ALT, aspartate aminotransferase (AST), bilirubin);
6. Normal renal function tests (creatinine, blood urea nitrogen (BUN), urinalysis);
7. Serum alpha-fetoprotein (AFP) negative.

Exclusion Criteria:

1. Pregnant (positive human chorionic gonadotropin (HCG) strip test)
2. Current or former diagnosis of cancer, with the exception of non-melanomatous skin cancer.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Excretion of sulforaphane and metabolites in urine | Consecutive overnight urine samples collected for the duration of the study (21 days)
  Levels of sulforaphane and its glutathione-conjugate derived metabolites will be measured in consecutive overnight urine samples

SECONDARY OUTCOMES:
Air pollution biomarkers in urine | Consecutive overnight urine samples collected for the duration of the study (21 days)
  Levels of benzene mercapturic acid excreted in urine

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Kensler, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Qidong Liver Cancer Institute, Qidong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon completion of biomarker analyses (January 2020)

REFERENCES:
- [Background] Egner PA, Chen JG, Zarth AT, Ng DK, Wang JB, Kensler KH, Jacobson LP, Munoz A, Johnson JL, Groopman JD, Fahey JW, Talalay P, Zhu J, Chen TY, Qian GS, Carmella SG, Hecht SS, Kensler TW. Rapid and sustainable detoxication of airborne pollutants by broccoli sprout beverage: results of a randomized clinical trial in China. Cancer Prev Res (Phila). 2014 Aug;7(8):813-823. doi: 10.1158/1940-6207.CAPR-14-0103. Epub 2014 Jun 9. PMID 24913818